CLINICAL TRIAL: NCT03377868
Title: Optic Coherence Tomography in Patients With Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Achraf Makki, Assistant professor, American University of Beirut Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IM.AS.01
Record Dates: First submitted 2017-12-06; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Respiratory Function Tests

STUDY DESIGN:
Intervention Model Description: Observational study of a cohort of patients with amyotrophic lateral sclerosis compared to a parallel cohort of healthy age and sex matched subjects
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with Amyotrophic lateral sclerosis (Other): Patients diagnosed with amyotrophic lateral sclerosis
  Interventions: Diagnostic Test: Optic coherence tomography; Diagnostic Test: Pulmonary function test
- Control (Other): Parallel cohort of healthy age and sex matched subjects
  Interventions: Diagnostic Test: Optic coherence tomography; Diagnostic Test: Pulmonary function test

INTERVENTIONS:
Diagnostic Test: Optic coherence tomography — Optic coherence tomography measures retinal layer thickness, macular volume , and cell inner plexiform layer.
Diagnostic Test: Pulmonary function test — Pulmonary function test measures forced vital capacity and forced expiratory volume in one second.

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is an adult-onset, devastating, neurodegenerative disease characterized by the loss of cortical, brain stem, and spinal motor neurons. Visual evoked potentials studies in patients with ALS suggest visual pathway involvement. Optic coherence tomography (OCT) is a non-invasive cross-sectional imaging modality measuring the optical reflections in biological tissues. The main objective of this observational cohort study is to explore the correlation between changes on OCT retinal parameters and and clinical disability as measured by the ALS Functional Rating Scale (ALS-FRS-r) in patients with ALS at baseline, 3 and 6 months. A secondary objective is to explore the correlation between changes in retinal OCT parameters and pulmonary function tests (FVC and FEV1) in this cohort of patients with ALS. A parallel cohort of healthy age and sex matched subjects will participate as controls to obtain reference values of their retinal layers' thickness at baseline, 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ALS according to the El Escorial criteria.
* Age 18 years to 80 years old
* Disease duration less than 36 months
* Patients logistically able to attend and be evaluated at baseline, 3 and 6 months

Exclusion Criteria:

* Patients with diabetes mellitus
* Patients with glaucoma, refractive errors of ± 6 diopters or more, or other ophthalmologic disorders such as media opacities that could interfere with retinal OCT assessment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-03 (Estimated); Primary Completion 2018-07-28 (Estimated); Study Completion 2018-09-28 (Estimated)

PRIMARY OUTCOMES:
Change in retinal layer thickness parameters over 3 and 6 months in ALS patients | 6 months
  Observing the change in retinal layers thickness parameters in micrometers in ALS patients from baseline to 3 and 6 months

SECONDARY OUTCOMES:
Comparison of changes in retinal layer thickness parameters over 3 and 6 months between ALS patients and their healthy controls | 6 month
  Comparison of changes in retinal layer thickness parameters over 3 and 6 months between ALS patients and their healthy controls in micrometers
Correlation between changes in retinal layers thickness and ALS-FRS scores in patients with ALS | 6 month
  Correlation between changes in retinal layers thickness in micrometers and ALS-FRS scores in ALS patients over 3 and 6 month
Correlation between changes in retinal layers thickness and Pulmonary function test parameters in ALS patients over 3 and 6 months | 6 month
  Correlation between changes in retinal layers thickness parameters in micrometers and changes in FEV1 in liters and FVC in liters on pulmonary function testing in patients with ALS over 3 and 6 month

REFERENCES:
- [Background] Calvo AC, Manzano R, Mendonca DM, Munoz MJ, Zaragoza P, Osta R. Amyotrophic lateral sclerosis: a focus on disease progression. Biomed Res Int. 2014;2014:925101. doi: 10.1155/2014/925101. Epub 2014 Aug 3. PMID 25157374
- [Background] Grosskreutz J, Kaufmann J, Fradrich J, Dengler R, Heinze HJ, Peschel T. Widespread sensorimotor and frontal cortical atrophy in Amyotrophic Lateral Sclerosis. BMC Neurol. 2006 Apr 25;6:17. doi: 10.1186/1471-2377-6-17. PMID 16638121
- [Background] Hammad M, Silva A, Glass J, Sladky JT, Benatar M. Clinical, electrophysiologic, and pathologic evidence for sensory abnormalities in ALS. Neurology. 2007 Dec 11;69(24):2236-42. doi: 10.1212/01.wnl.0000286948.99150.16. PMID 18071143
- [Background] Radtke RA, Erwin A, Erwin CW. Abnormal sensory evoked potentials in amyotrophic lateral sclerosis. Neurology. 1986 Jun;36(6):796-801. doi: 10.1212/wnl.36.6.796. PMID 3703285
- [Background] Munte TF, Troger MC, Nusser I, Wieringa BM, Johannes S, Matzke M, Dengler R. Alteration of early components of the visual evoked potential in amyotrophic lateral sclerosis. J Neurol. 1998 Apr;245(4):206-10. doi: 10.1007/s004150050206. PMID 9591221
- [Background] Moss HE, McCluskey L, Elman L, Hoskins K, Talman L, Grossman M, Balcer LJ, Galetta SL, Liu GT. Cross-sectional evaluation of clinical neuro-ophthalmic abnormalities in an amyotrophic lateral sclerosis population. J Neurol Sci. 2012 Mar 15;314(1-2):97-101. doi: 10.1016/j.jns.2011.10.016. Epub 2011 Dec 21. PMID 22192877
- [Background] Huang D, Swanson EA, Lin CP, Schuman JS, Stinson WG, Chang W, Hee MR, Flotte T, Gregory K, Puliafito CA, et al. Optical coherence tomography. Science. 1991 Nov 22;254(5035):1178-81. doi: 10.1126/science.1957169.
- [Background] Puliafito CA, Hee MR, Lin CP, Reichel E, Schuman JS, Duker JS, Izatt JA, Swanson EA, Fujimoto JG. Imaging of macular diseases with optical coherence tomography. Ophthalmology. 1995 Feb;102(2):217-29. doi: 10.1016/s0161-6420(95)31032-9. PMID 7862410
- [Background] Jimenez B, Ascaso FJ, Cristobal JA, Lopez del Val J. Development of a prediction formula of Parkinson disease severity by optical coherence tomography. Mov Disord. 2014 Jan;29(1):68-74. doi: 10.1002/mds.25747. Epub 2013 Nov 14. PMID 24458320
- [Background] Ascaso FJ, Cruz N, Modrego PJ, Lopez-Anton R, Santabarbara J, Pascual LF, Lobo A, Cristobal JA. Retinal alterations in mild cognitive impairment and Alzheimer's disease: an optical coherence tomography study. J Neurol. 2014 Aug;261(8):1522-30. doi: 10.1007/s00415-014-7374-z. Epub 2014 May 21. PMID 24846203
- [Background] Bertuzzi F, Suzani M, Tagliabue E, Cavaletti G, Angeli R, Balgera R, Rulli E, Ferrarese C, Miglior S. Diagnostic validity of optic disc and retinal nerve fiber layer evaluations in detecting structural changes after optic neuritis. Ophthalmology. 2010 Jun;117(6):1256-1264.e1. doi: 10.1016/j.ophtha.2010.02.024. Epub 2010 Apr 9. PMID 20381872
- [Background] Bennett JL, de Seze J, Lana-Peixoto M, Palace J, Waldman A, Schippling S, Tenembaum S, Banwell B, Greenberg B, Levy M, Fujihara K, Chan KH, Kim HJ, Asgari N, Sato DK, Saiz A, Wuerfel J, Zimmermann H, Green A, Villoslada P, Paul F; GJCF-ICC&BR. Neuromyelitis optica and multiple sclerosis: Seeing differences through optical coherence tomography. Mult Scler. 2015 May;21(6):678-88. doi: 10.1177/1352458514567216. Epub 2015 Feb 6. PMID 25662342
- [Background] Roth NM, Saidha S, Zimmermann H, Brandt AU, Oberwahrenbrock T, Maragakis NJ, Tumani H, Ludolph AC, Meyer T, Calabresi PA, Paul F. Optical coherence tomography does not support optic nerve involvement in amyotrophic lateral sclerosis. Eur J Neurol. 2013 Aug;20(8):1170-6. doi: 10.1111/ene.12146. Epub 2013 Apr 14. PMID 23582075
- [Background] Ringelstein M, Albrecht P, Sudmeyer M, Harmel J, Muller AK, Keser N, Finis D, Ferrea S, Guthoff R, Schnitzler A, Hartung HP, Methner A, Aktas O. Subtle retinal pathology in amyotrophic lateral sclerosis. Ann Clin Transl Neurol. 2014 Apr;1(4):290-7. doi: 10.1002/acn3.46. Epub 2014 Mar 11. PMID 25590041
- [Background] Simonett JM, Huang R, Siddique N, Farsiu S, Siddique T, Volpe NJ, Fawzi AA. Macular sub-layer thinning and association with pulmonary function tests in Amyotrophic Lateral Sclerosis. Sci Rep. 2016 Jul 7;6:29187. doi: 10.1038/srep29187. PMID 27383525
- [Background] Saidha S, Al-Louzi O, Ratchford JN, Bhargava P, Oh J, Newsome SD, Prince JL, Pham D, Roy S, van Zijl P, Balcer LJ, Frohman EM, Reich DS, Crainiceanu C, Calabresi PA. Optical coherence tomography reflects brain atrophy in multiple sclerosis: A four-year study. Ann Neurol. 2015 Nov;78(5):801-13. doi: 10.1002/ana.24487. Epub 2015 Oct 1. PMID 26190464